CLINICAL TRIAL: NCT05459636
Title: Time-Efficient Inspiratory Muscle Strength Training as a New Approach to Lower Blood Pressure, Improve Respiratory Function, and Reduce Exertional Dyspnea in Adults With Obesity
Brief Title: Inspiratory Muscle Strength Training in Adults With Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Joseph Watso, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00003098; K01HL160772 (NIH)
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High-resistance inspiratory muscle strength training (Active Comparator): Participants will perform high-resistance inspiratory muscle strength training on a daily basis for eight weeks using a handheld device that produces resistance that increases the effort of breathing in.
  Interventions: Device: High-resistance inspiratory muscle strength training
- Very-low resistance inspiratory muscle strength training (Sham Comparator): Participants will perform very-low-resistance inspiratory muscle strength training on a daily basis for eight weeks using a handheld device that produces resistance that increases the effort of breathing in.
  Interventions: Device: Very-low-resistance inspiratory muscle strength training

INTERVENTIONS:
Device: High-resistance inspiratory muscle strength training — Participants will perform high-resistance inspiratory muscle strength training on a daily basis for eight weeks using a handheld device that produces resistance that increases the effort of breathing in.
  Arms: High-resistance inspiratory muscle strength training
Device: Very-low-resistance inspiratory muscle strength training — Participants will perform very-low-resistance inspiratory muscle strength training on a daily basis for eight weeks using a handheld device that produces resistance that increases the effort of breathing in.
  Arms: Very-low resistance inspiratory muscle strength training

SUMMARY:
The purpose of this study is to determine whether inspiratory muscle strength training reduces blood pressure in adults with obesity.

DETAILED DESCRIPTION:
Obesity affects four-in-ten American adults and is associated with hypertension and greater all-cause mortality. Irrespective of weight loss, aerobic exercise reduces arterial blood pressure (BP) and improves cardiometabolic health. However, nearly half of adults with obesity do not perform aerobic exercise because of low leisure time availability and exertional dyspnea secondary to high chest wall mass-related inspiratory muscle dysfunction. In other clinical populations, emerging data demonstrates time-efficient high-resistance inspiratory muscle strength training (IMST) reduces BP and improves respiratory muscle function. Therefore, the investigators will determine whether eight weeks of daily high-resistance IMST reduces BP, improves respiratory muscle function, and concomitantly reduces exertional dyspnea in a randomized, double-blinded, sham-controlled (i.e., very low-resistance IMST) clinical trial among adults with obesity

ELIGIBILITY:
Inclusion Criteria:

- Body mass index 30 - 40 kg/m2

Exclusion Criteria:

* Not weight stable (<5% change in body mass over the past six months)
* Overt cardiovascular, neurological, renal, liver, and/or metabolic illness (e.g., diabetes mellitus)
* Current, or history of uncontrolled, Stage 2 hypertension (blood pressure >140 / 90 mmHg; anti-hypertensive medications are permitted)
* Diagnosed obstructive sleep apnea
* Previous bariatric surgery
* Diagnosis or signs (e.g., values below the lower limit of normal) of overt airway disease(s)
* Current or recent (regular use within the past 6 months) use of tobacco or nicotine products (e.g., cigarettes, vaping)
* Pregnant (self-reported and confirmed via urine pregnancy test), lactating (self-reported), or post-menopausal (self-reported) females
* Prisoners
* Per the POWERbreathe® company:

  * Patients who have undergone recent abdominal surgery and those with abdominal hernia.
  * Asthma patients who have a very low symptom perception and suffer from frequent, severe exacerbations or with an abnormally low perception of dyspnea.
  * If a patient is suffering from a ruptured eardrum or any other condition of the ear.
  * Patients with marked elevated left ventricular end-diastolic volume and pressure.
  * Patients with worsening heart failure signs and symptoms after training.
  * If an individual is suffering from a cold, sinusitis or respiratory tract infection, it is advised that they do not use the POWERbreathe device.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in laboratory-measured blood pressure | Up to 16 weeks
  Systolic and diastolic blood pressure measured in the laboratory

SECONDARY OUTCOMES:
Change in ambulatory blood pressure | Up to 16 weeks
  Systolic and diastolic blood pressure measured at home using an automated monitor
Change in inspiratory muscle strength | Up to 16 weeks
  Peak inspiratory pressure measured in the laboratory
Change in blood pressure reactivity during aerobic exercise | Up to 16 weeks
  Systolic and diastolic blood pressure measured in the laboratory at rest and during an incremental aerobic exercise test
Blood pressure during respiratory muscle testing | Up to 16 weeks
  Systolic and diastolic blood pressure measured in the laboratory at rest and during a respiratory muscle exercise test (eucapnic voluntary hyperpnea)

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with all HIPAA identifiers removed may be shared in future collaborative efforts pending appropriate data and/or material transfer agreement approvals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after completion of trial, indefinitely
Access Criteria: A formal plan identifying the intended use of the data and proper completion of appropriate data and/or material transfer agreement approvals with the study PI and their institution.